CLINICAL TRIAL: NCT00871143
Title: Efficacy of Cognitive Behaviour Therapy -v- Anxiety Management for Body Dysmorphic Disorder: a Randomised Controlled Trial
Brief Title: Cognitive Behaviour Therapy (CBT) for Body Dysmorphic Disorder (BDD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Psychiatry, London (Other)
Responsible Party: Principal Investigator, David Veale, Consultant Psychiatrist, Institute of Psychiatry, London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAXKAYR; 0 (Other: Institute of Psychiatry)
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Results first posted 2015-10-06 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-09

CONDITIONS: Body Dysmorphic Disorder
Keywords: CBT; BDD
MeSH Terms: conditions — Body Dysmorphic Disorders | interventions — 7,7'-dimethoxy-(4,4'-bi-1,3-benzodioxole)-5,5'-dicarboxylic acid dimethyl ester

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT specific for BDD (Experimental): This consisted of 12 wks of 1 hr sessions (1 per week).The consisted of engagement in a developmental understanding of the problem and setting up an alternative view of the problem. Imagery rescripting followed for past aversive memories that were associated with the onset (e.g. bullying). The behaviours were aimed at either (1) threat detection and monitoring or (2) preventing feared consequences by avoidance or (3) attempts to undo the appearance concerns. The therapist aimed to help individuals identify their beliefs about processes, conduct behavioural experiments that tested out their expectations and to gradually drop the safety-seeking behaviours and test out their fears.
  Interventions: Behavioral: CBT specific for BDD
- Non Specific CBT (Active Comparator): Anxiety Management treatment was provided once a week for 12 weeks, with each session lasting 1 hr. AM was planned to entail a therapeutic alliance, support and homework similar to the CBT group. The rationale provided was that when triggered, the person would experience a threat and negative thoughts about their appearance. This, in turn, would lead to physical symptoms of anxiety and magnify the perceived threat. The treatment consisted of (1) practising progressive muscle relaxation and breathing daily, (2) identifying triggers and physical symptoms associated with appearance-related anxiety and (3) utilising brief muscle relaxation and breathing techniques in trigger situations.
  Interventions: Behavioral: Non specific CBT

INTERVENTIONS:
Behavioral: CBT specific for BDD — This consisted of 12 wks of 1 hr sessions (1 per week).The consisted of engagement in a developmental understanding of the problem and setting up an alternative view of the problem. Imagery rescripting followed for past aversive memories that were associated with the onset (e.g. bullying). The behaviours were aimed at either (1) threat detection and monitoring or (2) preventing feared consequences by avoidance or (3) attempts to undo the appearance concerns. The therapist aimed to help individuals identify their beliefs about processes, conduct behavioural experiments that tested out their expectations and to gradually drop the safety-seeking behaviours and test out their fears.
  Arms: CBT specific for BDD
Behavioral: Non specific CBT — Anxiety Management treatment was provided once a week for 12 weeks, with each session lasting 1 hr. AM was planned to entail a therapeutic alliance, support and homework similar to the CBT group. The rationale provided was that when triggered, the person would experience a threat and negative thoughts about their appearance. This, in turn, would lead to physical symptoms of anxiety and magnify the perceived threat. The treatment consisted of (1) practising progressive muscle relaxation and breathing daily, (2) identifying triggers and physical symptoms associated with appearance-related anxiety and (3) utilising brief muscle relaxation and breathing techniques in trigger situations.
  Arms: Non Specific CBT

SUMMARY:
The aim of the research is to determine if Cognitive Behaviour Therapy (CBT) specific for BDD is more effective than a credible non-specific form of CBT for treating BDD and its delusional variant in adults aged 17 or over. This will be done in a single centre randomised controlled trial that compares specific CBT for BDD versus non-specific CBT over 12 weeks. The hypotheses to be tested are that: (1) specific CBT for BDD will be more effective than non-specific CBT at 12 weeks (2) Treatment effects from Specific CBT will be maintained at 1 month follow up. The main study end-point is at 12 weeks and the secondary end-point is at 1 month follow up. A secondary aim is to explore whether delusionality (insight) as measured by the Brown Assessment of Beliefs and co-morbid depressed mood predicts response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* BDD is the main psychological problem. We will use DSMIV criteria as BDD does not exist as a separate diagnosis in ICD10. They may have an additional diagnosis of Delusional Disorder when it refers to beliefs about being ugly or defective.
* They must have a total of 24 or more on the twelve-item YBOCS modified for BDD (Phillips et al., 1997).
* They may be of either gender but must be 17 years or above.
* They are willing to travel to the treatment centre for weekly sessions.
* They are wiling to complete regular questionnaires and be audiotaped for supervision and for listening to enhance their learning.
* They may be taking psychotropic medication so long as it is stabilised and there are no plans to increase the dose.

Exclusion Criteria:

* They have a current or past diagnosis of schizophrenia, bipolar affective disorder.
* They have current suicidal intent or severe self-neglect that requires hospitalisation.
* They have a current alcohol or substance dependence or anorexia nervosa or borderline personality disorder that requires treatment in its own right.
* They are currently receiving any other form of psychotherapy,
* They have received CBT for BDD in the past 6 months, which is judged as competently delivered and did not respond.
* They cannot speak sufficient English for CBT. (Assistance will be provided for those who speak English but are unable to read questionnaires).

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-04; Primary Completion 2011-05 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- South London and Maudsley NHS Trust, London, United Kingdom

REFERENCES:
- [Result] Veale D, Anson M, Miles S, Pieta M, Costa A, Ellison N. Efficacy of cognitive behaviour therapy versus anxiety management for body dysmorphic disorder: a randomised controlled trial. Psychother Psychosom. 2014;83(6):341-53. doi: 10.1159/000360740. Epub 2014 Oct 16. PMID 25323062

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: April 2009-March 2012. Single location: outpatient clinic at the Centre for Anxiety Disorders and Trauma at the Maudsley Hospital, London.
  Follow-ups: December 2009- September 2012. The trial ended when all participants had completed the follow-up.
  Last participant was recruited March 2012;last follow up was completed Sept 2012.
Pre-assignment Details: It was initially decided that 42 participants would be enrolled in the study (21 in each group), however in order to anticipate potential future drop outs, 46 participants were randomised into the 2 groups.
Groups:
- CBT Specific for BDD: CBT specific for BDD: Cognitive behaviour therapy (CBT) which is specific for BDD. A pilot study (Veale et al, 1996b) twelve years ago has demonstrated significant benefit of CBT over a waiting list. The mean reduction was about 50% on the primary outcome measure (YBOCS for BDD). This consisted of a reduction of 12 points and a standard deviation of 7 on the YBOCS for BDD and the treatment is now thought to be better than in 1996.
- Non Specific CBT: Non specific CBT: CBT which is not specific for BDD (stress management and cognitive restructuring) which has been shown to be a credible alternative psychological treatment to CBT in health anxiety. However in two pilot cases of BDD, the benefits of anxiety management were minimal with a reduction of between zero and 10% on the YBOCS for BDD. At the most this equates to a maximum of 3 points reduction.
Period: Overall Study
Arm/Group | CBT Specific for BDD | Non Specific CBT
Started | 21 | 25
Completed | 21 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Inclusion criteria:
  * Diagnosis of BDD according to the DSM-IV diagnostic criterion
  * Total of >24 on the Yale-Brown Obsessive Compulsive Scale modified for BDD
  * >18 years old
  * Willing to travel to the treatment centre for weekly sessions
  * Not on psychotropic medication or on a dose that's been stable for at least 12 weeks
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT Specific for BDD | Non Specific CBT | Total
Number analyzed (Participants) | 21 | 25 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 25 | 46
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 30.0 [24.5 to 37.5] | 29.0 [25.5 to 37.0] | 30.0 [25.0 to 36.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 16 | 21 | 37
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 21 | 25 | 46
Yale-Brown Obsessive Compulsive Scale modified for BDD (BDD-YBOCS) [Mean (Standard Deviation); unit: units on a scale] — This is a clinician-rated scale administered by a trained blinded assessor. The range is 0-48. Cronbach's α for the scale is 0.80. Response to treatment is defined as a 30% or greater decrease in the total BDD-YBOCS score, which best corresponded to 'much improved' on the Clinical Global Impression (CGI) scale. In the original validation study, this cutoff score produced 1 false negative (96% sensitivity), that is, 1 participant who was rated as much or very much improved on the CGI was not classified as a responder on the BDD-YBOCS using the 30% threshold.
  units on a scale | 35.48 (6.61) | 37.68 (4.77) | 36.58 (5.69)
Brown Assessment of Beliefs Scale (BABS) [Mean (Standard Deviation); unit: units on a scale] — BABS is a 7-item clinician scale rated by a blinded assessor to measure the strength of conviction in a belief (e.g. 'I am as ugly as the Elephant man'); each item is rated from 0 ('non-delusional belief, or least pathological') to 4 ('delusional belief, or most pathological') and the total scores range from 0 to 24; higher scores represent an increasing delusionality of beliefs; respondents are classified as having delusional BDD beliefs if their total score is 18 or more, and if they score 4 on the first item, indicating they are completely convinced that their belief is accurate.
  units on a scale | 18.24 (4.68) | 18.96 (4.14) | 18.60 (4.41)
Montgomery-Åsberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — MADRS is a 10-item clinician scale rated by a blinded assessor to measure symptoms of depression; each item is rated on a 7-point Likert scale from 0 (indicating 'normal' or 'no difficulties') to 6, and the range is 0-60; higher scores reflect a greater symptomatology; a MADRS total score of ≥ 25 is regarded as moderate, and of >31 as severe.
  units on a scale | 28.57 (10.69) | 30.04 (9.62) | 29.31 (10.16)
Appearance Anxiety Inventory (AAI) [Mean (Standard Deviation); unit: units on a scale] — The AAI is a 10- item self-report questionnaire for measuring the frequency of avoidance behaviour and threat-monitoring (e.g. checking, self-focussed attention) that are characteristic of a response to a distorted body image; each item is scored from 0 ('not at all') to 4 ('all the time'), and the range of the total scores is 0-40, with higher scores reflecting a greater frequency of the responses; the AAI has a Cronbach's α of 0.86.
  units on a scale | 26.89 (6.62) | 27.78 (7.03) | 27.335 (6.83)
Patient Health Questionnaire (PHQ)-9 [Mean (Standard Deviation); unit: units on a scale] — The PHQ is a 9-item self-report measure of depression; each item is scored from 0 ('not at all') to 3 ('nearly every day'),and the summed total score ranges from 0 to 27, with higher scores reflecting a greater symptomatology of depression; Cronbach's α for the scale is 0.89.
  units on a scale | 13.10 (6.50) | 13.60 (5.44) | 13.35 (5.97)
Generalised Anxiety Disorder (GAD)-7 [Mean (Standard Deviation); unit: units on a scale] — The GAD-7 is a 7-item self-report measure for symptoms of generalised anxiety; each item is scored from 0 to 3, and the summed total score ranges from 0 to 21, with higher scores reflecting a greater symptomatology; Cronbach's α for the measure is 0.92.
  units on a scale | 11.33 (6.32) | 13.09 (5.24) | 12.21 (5.78)
Body Image Quality of Life Inventory (BIQLI) [Mean (Standard Deviation); unit: units on a scale] — The BIQLI is a 19-item self-report scale that measures the impact of body image concerns on a broad range of life domains (e.g. sense of self, social functioning, sexuality, emotional well-being, exercise and grooming); the BIQLI is scored as the average numeric score of all the items from -3 ('very negative effect') to +3 ('very positive effect'); Cronbach's α for the scale is 0.95.
  units on a scale | -1.97 (0.56) | -1.68 (1.04) | -1.83 (0.80)

OUTCOME MEASURES:

1. Primary Outcome: Yale Brown Obsessive Compulsive Scale (Modified for BDD) (BDD -YBOCS) (Phillips et al., 1997)
Description: This is a clinician-rated scale administered by a trained blinded assessor. The range is 0-48. Cronbach's α for the scale is 0.80. Response to treatment is defined as a 30% or greater decrease in the total BDD-YBOCS score, which best corresponded to 'much improved' on the Clinical Global Impression (CGI) scale. In the original validation study, this cutoff score produced 1 false negative (96% sensitivity), that is, 1 participant who was rated as much or very much improved on the CGI was not classified as a responder on the BDD-YBOCS using the 30% threshold.
Time Frame: 12 weeks, 1 month post treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Non Specific CBT: Non specific CBT: CBT which is not specific for BDD (stress management and cognitive restructuring) which has been shown to be a credible alternative psychological treatment to CBT in health anxiety. However in two pilot cases of BDD, the benefits were minimal with a reduction of between zero and 10% on the YBOCS for BDD. At the most this equates to a maximum of 3 points reduction.
Arm/Group | CBT Specific for BDD | Non Specific CBT
Number analyzed (Participants) | 21 | 25
units on a scale
  12 weeks | 23.47 (11.23) | 32.87 (7.45)
  1 month | 21.37 (12.42) | 33.30 (8.72)
Statistical Analysis 1: Comparison: CBT Specific for BDD; Linear mixed models were conducted to determine the predictive value of treatment group and/or time on the outcome variable scores; Test type: Superiority or Other; p < .001, Mixed Models Analysis — An alpha level of .05 (two-sided) was set
Statistical Analysis 2: Comparison: CBT Specific for BDD; Investigating the difference in BDD YBOCS score between baseline and week 12; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferroni correction was used to decrease the risk of type I error
Statistical Analysis 3: Comparison: CBT Specific for BDD; Investigating the difference in BDD YBOCS score between between baseline and 1 month follow up; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferroni corrections were used to reduce risk of Type 1 error
Statistical Analysis 4: Comparison: Non Specific CBT; Investigating the difference in BDD YBOCS score between baseline and week 12; Test type: Superiority or Other; p < .01, t-test, 2 sided — Bonferroni correction was used to decrease the risk of type I error
Statistical Analysis 5: Comparison: Non Specific CBT; Investigating the difference in BDD YBOCS score between baseline and 1 month follow up; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — Bonferroni correction was used to decrease risk of type I error

2. Secondary Outcome: Brown Assessment of Beliefs to Measure the Strength of Conviction in Beliefs About Being Ugly (Eisen et al., 1998)
Description: BABS is a 7-item clinician scale rated by a blinded assessor to measure the strength of conviction in a belief (e.g. 'I am as ugly as the Elephant man'); each item is rated from 0 ('non-delusional belief, or least pathological') to 4 ('delusional belief, or most pathological') and the total scores range from 0 to 24; higher scores represent an increasing delusionality of beliefs; respondents are classified as having delusional BDD beliefs if their total score is 18 or more, and if they score 4 on the first item, indicating they are completely convinced that their belief is accurate.
Time Frame: 12 weeks, 1 month post treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT Specific for BDD | Non Specific CBT
Number analyzed (Participants) | 21 | 25
units on a scale
  12 week | 12.75 (8.11) | 17.92 (5.42)
  1 month | 10.28 (7.41) | 18.88 (4.62)
Statistical Analysis 1: Comparison: CBT Specific for BDD vs Non Specific CBT; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .05, Mixed Models Analysis — An alpha level of .05 was set (two-sided)
Statistical Analysis 2: Comparison: CBT Specific for BDD; T-tests were used to investigate significant differences between baseline and 12 week measures; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — Bonferroni correction was used to decrease the risk of type I error
Statistical Analysis 3: Comparison: CBT Specific for BDD; T-tests were used to investigate significant differences between baseline and 1 month follow up; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Bonferroni corrections were implemented to adjust for type I error
Statistical Analysis 4: Comparison: Non Specific CBT; T-tests were used to investigate significant differences between baseline and 12 week assessment measures and baseline and 1 month follow up measures; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Bonferroni correction was used to decrease the risk of type I error
Statistical Analysis 5: Comparison: Non Specific CBT; T-tests were used to investigate significant differences between baseline and 1 month follow up measures; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Bonferroni corrections were used to reduce risk of type I error

3. Secondary Outcome: Montgomery Asberg Depression Rating Scale (Montgomery and Asberg, 1979).
Description: MADRS is a 10-item clinician scale rated by a blinded assessor to measure symptoms of depression; each item is rated on a 7-point Likert scale from 0 (indicating 'normal' or 'no difficulties') to 6, and the range is 0-60; higher scores reflect a greater symptomatology; a MADRS total score of ≥ 25 is regarded as moderate, and of >31 as severe.
Time Frame: 12 weeks, 1 month post treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT Specific for BDD | Non Specific CBT
Number analyzed (Participants) | 21 | 25
units on a scale
  12 week | 21.71 (11.20) | 25.98 (10.80)
  1 month | 20.40 (13.14) | 28.63 (13.32)
Statistical Analysis 1: Comparison: CBT Specific for BDD vs Non Specific CBT; A Linear mixed model was conducted to determine the predictive value of treatment group and/or time on the outcome variable MADRS scores; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis — An alpha level of .05 was set (two-sided)
Statistical Analysis 2: Comparison: CBT Specific for BDD; Investigating the difference in MADRS score between baseline and week 12; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — Bonferroni correction was used to decrease the risk of type I error
Statistical Analysis 3: Comparison: CBT Specific for BDD; Investigating the difference in MADRS score between baseline and 1 month follow up; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Bonferonni corrections used to reduce risk of type I error
Statistical Analysis 4: Comparison: Non Specific CBT; Investigating the difference in MADRS score between baseline and week 12; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Bonferroni correction was used to decrease the risk of type I error
Statistical Analysis 5: Comparison: Non Specific CBT; Investigating the difference in MADRS score between baseline and 1 month follow up; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Bonferroni corrections used to decrease risk of type I error

4. Secondary Outcome: Appearance Anxiety Inventory (AAI)
Description: The AAI is a 10- item self-report questionnaire for measuring the frequency of avoidance behaviour and threat-monitoring (e.g. checking, self-focussed attention) that are characteristic of a response to a distorted body image; each item is scored from 0 ('not at all') to 4 ('all the time'), and the range of the total scores is 0-40, with higher scores reflecting a greater frequency of the responses; the AAI has a Cronbach's α of 0.86.
Time Frame: 12 weeks, 1 month post treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT Specific for BDD | Non Specific CBT
Number analyzed (Participants) | 21 | 25
units on a scale
  12 week | 14.61 (9.20) | 23.37 (8.29)
  1 month | 14.16 (9.53) | 23.21 (8.86)
Statistical Analysis 1: Comparison: CBT Specific for BDD vs Non Specific CBT; Linear mixed models were conducted to determine the predictive value of treatment group and/or time on the outcome variable of AAI scores; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — An alpha level of .05 (two-sided) was set
Statistical Analysis 2: Comparison: CBT Specific for BDD; Repeated- measures t tests were used to determine where significant differences in AAI scores occurred from baseline to 12 week; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Bonferroni corrections were applied to decrease the risk of type I error
Statistical Analysis 3: Comparison: CBT Specific for BDD; Repeated- measures t tests were used to determine where significant differences in AAI scores occurred from baseline to 2 month follow up; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Bonferroni corrections were used to reduce risk of type 1 error
Statistical Analysis 4: Comparison: Non Specific CBT; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — Bonferroni Correction was used in an attempt to reduce risk of type I error
Statistical Analysis 5: Comparison: Non Specific CBT; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Bonferroni corrections were used to adjust for type 1 error

5. Secondary Outcome: Patient Health Questionnaire (PHQ)-9
Description: The PHQ is a 9-item self-report measure of depression; each item is scored from 0 ('not at all') to 3 ('nearly every day'),and the summed total score ranges from 0 to 27, with higher scores reflecting a greater symptomatology of depression; Cronbach's α for the scale is 0.89.
Time Frame: 12 weeks, 1 month post treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT Specific for BDD | Non Specific CBT
Number analyzed (Participants) | 21 | 25
units on a scale
  12 week | 9.12 (7.01) | 13.28 (7.18)
  1 month | 9.41 (6.67) | 15.79 (7.05)
Statistical Analysis 1: Comparison: CBT Specific for BDD vs Non Specific CBT; Linear mixed models were conducted to determine the predictive value of treatment group and/or time on the PHQ-9 score; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis — An alpha level of .05 was set (two-sided)
Statistical Analysis 2: Comparison: CBT Specific for BDD; Repeated- measures t tests were used to determine where significant differences occurred from baseline to end of treatment (12 weeks); Test type: Superiority or Other; p < 0.05, t-test, 2 sided — Where more than 1 t test had been conducted on each variable, a Bonferroni correction was used to decrease the risk of type I error
Statistical Analysis 3: Comparison: CBT Specific for BDD; Repeated- measures t tests were used to determine where significant differences occurred from baseline to 2 month follow up; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Bonferroni corrections were used to reduce risk of type I error
Statistical Analysis 4: Comparison: Non Specific CBT; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — A Bonferroni correction was used to decrease the risk of type I error
Statistical Analysis 5: Comparison: Non Specific CBT; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Bonferroni corrections were used to reduce risk of type I error

6. Secondary Outcome: Generalised Anxiety Disorder (GAD)-7
Description: The GAD-7 is a 7-item self-report measure for symptoms of generalised anxiety; each item is scored from 0 to 3, and the summed total score ranges from 0 to 21, with higher scores reflecting a greater symptomatology; Cronbach's α for the measure is 0.92.
Time Frame: 12 weeks,1 month post treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT Specific for BDD | Non Specific CBT
Number analyzed (Participants) | 21 | 25
units on a scale
  12 week | 7.00 (6.02) | 11.59 (5.89)
  1 month | 8.53 (6.60) | 13.22 (5.45)
Statistical Analysis 1: Comparison: CBT Specific for BDD vs Non Specific CBT; Linear mixed models were conducted to determine the predictive value of treatment group and/or time on GAD-7 scores; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — An alpha level of .05 was set (two-sided)
Statistical Analysis 2: Comparison: CBT Specific for BDD; Repeated- measures t tests were used to determine where significant differences occurred from baseline to 12 week assessment; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — A Bonferroni correction was used to decrease the risk of type I error
Statistical Analysis 3: Comparison: CBT Specific for BDD; Repeated- measures t tests were used to determine where significant differences occurred from baseline to 2 month follow up assessment; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Bonferroni corrections were implemented to reduce the risk of type I error
Statistical Analysis 4: Comparison: Non Specific CBT; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — A Bonferroni correction was used to decrease the risk of type I error
Statistical Analysis 5: Comparison: Non Specific CBT; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Bonferroni corrections were used to reduce risk of type I error

7. Secondary Outcome: Body Image Quality of Life Inventory (BIQLI)
Description: The BIQLI is a 19-item self-report scale that measures the impact of body image concerns on a broad range of life domains (e.g. sense of self, social functioning, sexuality, emotional well-being, exercise and grooming); the BIQLI is scored as the average numeric score of all the items from -3 ('very negative effect') to +3 ('very positive effect'); Cronbach's α for the scale is 0.95.
Time Frame: 12 weeks, 1 month post treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT Specific for BDD | Non Specific CBT
Number analyzed (Participants) | 21 | 25
units on a scale
  12 week | -1.43 (0.85) | -2.04 (0.71)
  1 month | -1.29 (0.92) | -1.95 (0.81)
Statistical Analysis 1: Comparison: CBT Specific for BDD vs Non Specific CBT; Linear mixed models were conducted to determine the predictive value of treatment group and/or time on BIQLI scores; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — An alpha level of .05 was set (two-sided)
Statistical Analysis 2: Comparison: CBT Specific for BDD; Repeated-measures t tests were then used to determine where significant differences in BIQLI occurred between baseline and end of treatment (12 weeks); Test type: Superiority or Other; p < 0.05, t-test, 2 sided — A Bonferroni correction was used to decrease the risk of type I error
Statistical Analysis 3: Comparison: CBT Specific for BDD; Repeated-measures t tests were then used to determine where significant differences in BIQLI occurred between baseline and 1 month follow up; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — Bonferroni corrections were used to reduce risk of type 1 error
Statistical Analysis 4: Comparison: Non Specific CBT; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — A Bonferroni correction was used to decrease the risk of type I error
Statistical Analysis 5: Comparison: Non Specific CBT; [analysis description as in outcome 7, analysis 3]; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Bonferroni corrections were used

ADVERSE EVENTS:
Time Frame: Data on adverse events was not collected or assessed for this study.
Description: Data on adverse events was not collected or assessed for this study.
Arm/Group | CBT Specific for BDD | Non Specific CBT
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Small sample size: may have led to difficulty in identifying predictors of outcome.

Investigator bias: but testing blinding would be biased as it may be influenced by her rating of the outcome.

Treatment too brief to achieve sig. changes in BDD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes